CLINICAL TRIAL: NCT06619977
Title: Analgesia Nociception Index (ANI) for Guiding Intraoperative Opioid Administration During Living Donor Liver Resection and Its Impact on Postoperative Nausea and Vomiting
Brief Title: ANI-Guided Fentanyl Infusion During Living Donor Liver Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Nazarii Mysynchuk, MD, Bogomolets National Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 187
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-09

CONDITIONS: No Disease or Condition is Being Studied

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard practice retrospective group (No Intervention): Patients undergoing living liver donor resections with general anesthesia without ANI monitoring.
- ANI guided group (Experimental): Patients undergoing living liver donor resections with general anesthesia with ANI nociception monitoring.
  Interventions: Device: Analgesia nociception monitoring (ANI)

INTERVENTIONS:
Device: Analgesia nociception monitoring (ANI) — Analgesia nociception index (ANI; MetroDoloris Medical Systems, Lille, France) is a noninvasive tool for monitoring the intraoperative state of the autonomic nervous system, in particular - the parasympathetic nervous system. The ANI algorithm uses data from one lead ECG trace. Heart rate variability, or the beat-to-beat alterations in heart rate, is a well-known and recognised noninvasive indicator of autonomic nervous system activity.
  Arms: ANI guided group

SUMMARY:
Thу goal of this study was to learn whether intraoperative analgesia nociception monitoring (ANI) could be beneficial during intraoperative monitoring for patients undergoing living donor liver resections. The main questions it aims to answer are:

* Could it impact the average dose of intraoperative fentanyl used?
* Could it impact the occurrence of postoperative nausea and vomiting?

Patients who were included in this study underwent living liver donor resections with fentanyl infusion and thoracic epidural analgesia. Two groups of patients were analysed - the ANI group (n = 24), in which fentanyl dose was adjusted with ANI monitoring, and the retrospective control group (n = 25) with a standard practice without ANI monitoring.

DETAILED DESCRIPTION:
Monitoring nociception accurately during general anaesthesia has presented a long-standing difficulty. Typically, anaesthesiologists rely on changes in the autonomic nervous system, such as heart rate, blood pressure, and sweating, to help determine the need for pain relief medication. Analgesia nociception index (ANI) is a noninvasive tool for monitoring the intraoperative state of the autonomic nervous system, particularly the parasympathetic nervous system.

During the long-lasting high nociceptive surgery, the infusion of fentanyl was used at our institution. Opioids can lead to postoperative nausea, vomiting, and other complications when an overdose occurs. Fentanyl dosage changes significantly after hours of infusion due to context-sensitive halftime. It is practically impossible to adjust an infusion dose with the subjective evaluation of standard monitoring, such as heart rate and blood pressure. Doses of opioids that we use in our daily practice, e.g. mcg.kg-1, are unpredictable and vary between individuals due to pharmacogenetics and pharmacokinetic reasons. The best method to exclude pharmacokinetic peculiarities and predict the subsequent dose is to directly measure analgesic agents' concentration in the blood, though it is practically impossible. This study aimed to assess whether intraoperative analgesia nociception monitoring (ANI) could have an impact on the average intraoperative dose of fentanyl and on the occurrence of postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients, 18 - 60 years old, undergoing living donor liver resections with general anaesthesia with sevoflurane, thoracic epidural analgesia and fentanyl on infusion. ASA I, II

Exclusion Criteria:

* patients with cardiac arrhythmia (atrial fibrillation, frequent extrasystoles - more than one extrasystole in 30 seconds), total intravenous anaesthesia with propofol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Postoperative Nausea and Vomiting | from enrollment to the first 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Iurii Kuchyn, Professor of Anaesthesiology, Study Director — Bogomolets National Medical University, Kyiv, Ukraine
Locations (1):
- Universal Clinic Oberig, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No
Due to the institutional policy, the IPD will not be shared.